CLINICAL TRIAL: NCT07025642
Title: Outcome of Different Treatments of Overactive Bladder in Taiwan
Brief Title: Comparing Treatments for Overactive Bladder in Taiwan: A Study of Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, Head of administration, Mackay Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22MMHIS039e
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; mirabegron; Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- solifenacin (Experimental): oral solifenacin
  Interventions: Drug: Urodynamic evaluation before and after solifenacin treatment.
- mirabegron (Experimental): oral mirabegron
  Interventions: Drug: Urodynamic evaluation before and after mirabegron treatment.
- Solifenacin + mirabegron (Experimental): oral Solifenacin and mirabegron
  Interventions: Drug: Urodynamic evaluation before and after combined treatment with solifenacin and mirabegron.
- Botox (Experimental): Botox injection
  Interventions: Drug: Urodynamic evaluation before and after Botulinum toxin (Botox) injection.

INTERVENTIONS:
Drug: Urodynamic evaluation before and after solifenacin treatment. — Cystometry performed at 1 month before and 1, 6 months following/after treatments will be analyzed.
  Arms: solifenacin
Drug: Urodynamic evaluation before and after mirabegron treatment. — Cystometry performed at 1 month before and 1, 6 months following/after treatments will be analyzed.
  Arms: mirabegron
Drug: Urodynamic evaluation before and after combined treatment with solifenacin and mirabegron. — Cystometry performed at 1 month before and 1, 6 months following/after treatments will be analyzed.
  Arms: Solifenacin + mirabegron
Drug: Urodynamic evaluation before and after Botulinum toxin (Botox) injection. — Cystometry performed at 1 month before and 1, 6 months following/after treatments will be analyzed.
  Arms: Botox

SUMMARY:
Overactive bladder (OAB) syndrome is a prevalent condition that significantly impairs patients' quality of life. Standard therapeutic strategies include oral antimuscarinics (e.g., solifenacin), beta-3 adrenergic agonists (e.g., mirabegron), and intradetrusor injection of botulinum neurotoxin type A (BoNTA). Despite their clinical utility, these treatments share a common mechanism of action: suppression of detrusor muscle contractility. However, it remains unclear whether such suppression translates to a reduction in the overall mechanical work output of the bladder during micturition.

To address this question, our research proposes to assess how mirabegron, solifenacin, and BoNTA influence bladder function from a thermodynamic perspective. We will apply pressure-volume analysis (PVA), a methodology traditionally used in cardiac physiology, to quantify the mechanical work performed by the bladder per voiding cycle. This approach enables a direct measurement of the energy expenditure required for bladder emptying, offering insights beyond standard urodynamic parameters.

Furthermore, emerging data suggest BoNTA may exert additional effects beyond parasympathetic inhibition. Specifically, recent studies have demonstrated that BoNTA also inhibits norepinephrine release from sympathetic hypogastric nerve terminals. Since modulation of sympathetic activity-particularly via the hypogastric nerve-has been implicated in regulating bladder compliance and storage function, we hypothesize that BoNTA may influence bladder compliance through this secondary mechanism. To explore this, we will employ volume-pressure analysis (also abbreviated as PVA), which graphically represents the dynamic relationship between bladder volume and pressure throughout voiding cycles, thus capturing real-time changes in compliance.

Comparative studies of mirabegron, solifenacin, and BoNTA will allow us to differentiate their respective impacts on bladder work and compliance. Mirabegron, which selectively activates beta-3 adrenergic receptors, has minimal influence on overall sympathetic tone. In contrast, solifenacin not only antagonizes muscarinic receptors but may also indirectly potentiate sympathetic tone by reducing parasympathetic influence. BoNTA, with its dual action on both autonomic pathways, provides a unique model to dissect these neural mechanisms.

To extend our findings from clinical observations to preclinical validation, we aim to develop and utilize a spinal cord injury (SCI) rat model that recapitulates the bladder dysfunction observed in neurogenic detrusor overactivity (NDO)-a condition for which mirabegron, solifenacin, and BoNTA are also commonly prescribed. By applying both thermodynamic and compliance-focused PVA techniques in this animal model, we seek to construct a foundational database characterizing how these drugs modulate bladder function in a controlled, reproducible setting.

In summary, this project integrates a novel application of pressure- and volume-based analyses to quantify the mechanical and compliance-related effects of established OAB therapies in both human patients and a translational animal model. The findings will provide new mechanistic insights into how these treatments alter bladder physiology, potentially guiding future therapeutic strategies and optimizing drug selection for individualized patient care.

DETAILED DESCRIPTION:
BACKGROUND:

Year 1. Overactive bladder (OAB) syndrome remarkably places a burden on patients' quality of life. Given options for OAB therapies, namely oral anti-muscarinics, oral beta-3 agonists, and intra-detrusor botulinum neurotoxin type A (BoNTA) injection, involve trimming down of detrusor contractility, we wonder, if these modalities would diminish thermodynamic work performed by bladder. For this purpose, the impact of mirabgreon, solifenacin, and BoTNA on the work expenditure of bladder of OAB patients will be investigated using pressure-volume analysis (PVA), a protocol that thermodynamically quantifies work done by the bladder per voiding cycle.

Year 2. In addition to the well-established action, i.e., to impede acetylcholine release from the parasympathetic pelvic nerve, BoNTA also inhibits norepinephrine release from the ending of sympathetic hypogastric nerve. As a very recent work has linked adapted hypogastric tone to bladder compliance increment in patients with stress urinary incontinence, we wonder if via altering the activity of hypogastric nerve, intra-detrusor BoNTA injection would modify compliance to impact storage function of the bladder. Hence, effects of mirabgreon (a drug barely affecting sympathetic tone), solifenacin (a drug potentiating sympathetic tone), and BoTNA on the compliance dynamics of OAB patients' bladder will be investigated using volume-pressure analysis (PVA), a protocol that graphically illustrate compliance dynamics of voiding cycles.

YEAR 3: Developing an animal model available for testing pharmacological and side effects of mirabgreon, solifenacin, and BoTNA would offer a platform bridging preclinical experiments to clinical trial. Because above therapies are also prescribed in the therapy for neurogenic detrusor overactivity (NDO) patients; moreover, spinal cord injury (SCI) has been well-accepted as an animal model mimicking the condition of NDO. We therefore, aim to establish database of the impact of mirabgreon, solifenacin, and BoTNA on the thermodynamic work and compliance dynamics of NDO-like rats using the SCI model.

ELIGIBILITY:
Inclusion Criteria:

- female overactive bladder

Exclusion Criteria:

* DM, CVA, other medical problems

Ages: 30 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
pressure-volume analysis | within a voiding cycle (a cycle is about 30 to 60 minutes) 1-4 weeks before and 6-12 month after the operation
  urine leakage.
volume-pressure analysis | within a voiding cycle (a cycle is about 30 to 60 minutes) 1-4 weeks before and 6-12 month after the operation
  urine leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Shing Leu, M.D., Study Chair — Department of Ear, Nose, and Throat, MacKay Memorial Hospital, Taipei, Taiwan
Locations (1):
- Department of Obstetrics and Gynecology, New Taipei City, Taiwan